CLINICAL TRIAL: NCT05330858
Title: The Relative Bioavailability of an ESK-001 Tablet Versus Liquid Formulation, and the Effect of Food or Gastric Acid Reduction on the Pharmacokinetics of ESK-001 in Healthy Participants
Brief Title: Relative Bioavailability of ESK-001 Tablet Versus Liquid in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alumis Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ESK-001-002
Record Dates: First submitted 2022-03-30; First posted 2022-04-15 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ESK-001 Liquid (Experimental): ESK-001 administered as an oral liquid
  Interventions: Drug: ESK-001
- ESK-001 Tablet Fasted (Experimental): ESK-001 administered as an oral tablet in the fasted state
  Interventions: Drug: ESK-001
- ESK-001 Tablet Fed (Experimental): ESK-001 administered as an oral tablet in the fed state
  Interventions: Drug: ESK-001
- ESK-001 and Rabeprazole (Experimental): ESK-001 administered as an oral tablet with rabeprazole
  Interventions: Drug: ESK-001; Drug: Rabeprazole

INTERVENTIONS:
Drug: ESK-001 — Oral tablet or liquid
Drug: Rabeprazole — Oral Tablet
  Arms: ESK-001 and Rabeprazole

SUMMARY:
This is a single-center, in-house, open-label, crossover study in 15 healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Men and woman age 18-60
* Able to provide written informed consent
* Females can not be pregnant or lactating

Exclusion Criteria:

* Prior exposure to ESK-001
* History of malignancy within the last 10 years
* Positive for HIV, Hepatitis B or C
* History of tuberculosis
* Positive test for alcohol or drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Assess the PK parameters of ESK-001 via time of maximum plasma concentration (Tmax) | 18 Days
  Relative bioavailability and food effect assessment via collection and comparison of PK plasma samples between dosing arms
Assess the PK parameters of ESK-001 via maximum plasma concentration (Cmax) | 18 Days
  Relative bioavailability and food effect assessment via collection and comparison of PK plasma samples between dosing arms
Assess the PK parameters of ESK-001 via area under the concentration time curve (AUC) | 18 Days
  Relative bioavailability and food effect assessment via collection and comparison of PK plasma samples between dosing arms

SECONDARY OUTCOMES:
Assess the Incidence of Treatment Emergent Adverse Events of ESK-001 | 25 Days
  Collection and review of incidence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Alumis Central Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No